CLINICAL TRIAL: NCT06336902
Title: A Phase Ib Study of Botensilimab Plus Balstilimab and Fasting-Mimicking Diet (FMD) Plus Vitamin C in Patients With KRAS-Mutant Metastatic Colorectal Cancer
Brief Title: Botensilimab Plus Balstilimab and Fasting Mimicking Diet Plus Vitamin C for Patients With KRAS-Mutant Metastatic Colorectal Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3C-23-11; NCI-2024-01368 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 3C-23-11 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2024-03-21; First posted 2024-03-29 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Colorectal Adenocarcinoma; Stage IV Colorectal Cancer AJCC v8
MeSH Terms: conditions — Colorectal Neoplasms | interventions — balstilimab; Specimen Handling; Diet Therapy; Magnetic Resonance Spectroscopy; Ascorbic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (botensilimab, balstilimab, FMD, vitamin C) (Experimental): Patients receive botensilimab IV over 30 minutes on day 1 of each cycle for up to 4 cycles. Patients receive balstilimab IV over 30 minutes and vitamin C IV over 30 minutes on days 1, 15 and 29 of each cycle. Patients undergo a FMD on days -4 to -1 of each cycle. Cycles repeat every 42 days for up to 2 years in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo blood sample collection, CT scans and MRI throughout the study.
  Interventions: Biological: Balstilimab; Procedure: Biospecimen Collection; Biological: Botensilimab; Procedure: Computed Tomography; Other: Dietary Intervention; Procedure: Magnetic Resonance Imaging; Dietary Supplement: Vitamin C

INTERVENTIONS:
Biological: Balstilimab — Given IV
  Other Names: AGEN 2034; AGEN-2034; AGEN2034
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Biological: Botensilimab — Given IV
  Other Names: AGEN 1181; AGEN-1181; AGEN1181; Anti-CTLA-4 Monoclonal Antibody AGEN1181
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Other: Dietary Intervention — Undergo FMD
  Other Names: Dietary Modification; intervention, dietary; Nutrition Intervention; Nutrition Interventions; Nutritional Interventions
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Dietary Supplement: Vitamin C — Given IV

SUMMARY:
This phase Ib trial tests the safety, side effects, and effectiveness of botensilimab, and balstilimab in combination with a fasting mimicking diet and high dose vitamin C in treating patients with KRAS-mutant metastatic colorectal cancer. Botensilimab and balstilimab are monoclonal antibodies that may interfere with the ability of tumor cells to grow and spread. KRAS is protein found on some tumor cells that is involved in the growth of tumor cells. KRAS mutant cells have been found to be more sensitive to vitamin C induced growth suppression in the presence of low-sugar (glucose). A fasting mimicking diet, a plant-based, calorie reduced, low-sugar diet alternating with refeeding periods, may positively change the way the body responds to cancer treatment. Vitamin C is a nutrient that the body needs in small amounts to function and stay healthy. It is an antioxidant that that can help prevent cell damage and may block growth and spread of tumor cells. Botensilimab and balstilimab in combination with a fasting mimicking diet and high dose vitamin C may be safe, tolerable and effective in treating patients with KRAS-mutant metastatic colorectal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the feasibility of the fasting mimicking diet (FMD) when combined with vitamin C and botensilimab plus balstilimab by determining the proportion of patients who adhere to the FMD ≥ 75% of the designated days and receive all doses of botensilimab, balstilimab and Vitamin C for at least any two cycles of therapy.

II. To characterize the safety and tolerability of FMD and vitamin C when combined with botensilimab and balstilimab by assessing any grade toxicities per Common Terminology Criteria for Adverse Events (CTCAE) 5.0.

SECONDARY OBJECTIVES:

I. To obtain a preliminary assessment of anti-tumor activity of botensilimab plus balstilimab and FMD plus vitamin C by determining the overall response rate using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.

II. To estimate the progression-free and overall survival in patients with KRAS-mutant colorectal cancer (CRC) receiving botensilimab plus balstilimab and FMD plus vitamin C.

EXPLORATORY OBJECTIVES:

I. To characterize circulating tumor deoxyribonucleic acid (ctDNA) and ctDNA methylation (TET, Wnt, JAK/STAT, PI3K/AKT, CXCR, ALDH, AMPK) profiles at baseline, on treatment and at disease progression.

II. To examine metabolomic markers (IGF-1, GAPDH, DHA, GLUT-1, iron signaling) at baseline, on treatment and at disease progression.

OUTLINE:

Patients receive botensilimab intravenously (IV) over 30 minutes on day 1 of each cycle for up to 4 cycles. Patients receive balstilimab IV over 30 minutes and vitamin C IV over 30 minutes on days 1, 15 and 29 of each cycle. Patients undergo a FMD on days -4 to -1 of each cycle. Cycles repeat every 42 days for up to 2 years in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo blood sample collection, computed tomography (CT) scans and magnetic resonance imaging (MRI) throughout the study.

After completion of study intervention, patients are followed up at 30 days and every 3 months for up to 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed microsatellite stable (MSS) metastatic colorectal adenocarcinoma with any KRAS mutation (as determined by a Clinical Laboratory Improvement Act [CLIA]-certified lab), including metastases to liver, lung, etc.
* Disease progression, intolerance or contraindication to a fluoropyrimidine, oxaliplatin, irinotecan
* ≥ 18 years of age
* Performance status Eastern Cooperative Oncology Group (ECOG) 0-1
* Estimated life expectancy ≥ 3 months
* Body mass index (BMI) ≥ 18.5
* Absolute neutrophil count ≥ 1,500/mcL
* Hemoglobin ≥ 8.0 g/dL
* Platelets ≥ 75,000/mcL
* Total bilirubin ≤ 1.5 x upper limit of normal (ULN) (for patients with Gilbert syndrome ≤ 3.0 x ULN)
* Aspartate aminotransferase (AST) / alanine aminotransferase (ALT) ≤ 3 x ULN
* Creatinine ≤ 1.5 x ULN
* Measurable disease as defined by RECIST 1.1
* No history of prior or current malignancy that requires active treatment
* Female patients of childbearing potential must be willing to use highly effective contraceptive measures starting with the Screening visit through 90 days after last dose of study treatment.

Note: Abstinence is acceptable if this is the established and preferred contraception for the patient

* Female patients of childbearing potential must have a negative serum pregnancy test at screening (within 72 hours of first dose of study medication). Non-childbearing potential is defined as 1 of the following:

  * ≥ 45 years of age and has not had menses for > 1 year
  * Amenorrheic for > 2 years without a hysterectomy and/or oophorectomy and follicle stimulating hormone value in the postmenopausal range upon pretrial (screening) evaluation
  * Status is post-hysterectomy, -oophorectomy, or -tubal ligation
* Male patients with a female partner(s) of childbearing potential must agree to use highly effective contraceptive measures throughout the trial starting with the Screening visit through 90 days after the last dose of study treatment is received. Males with pregnant partners must agree to use a condom; no additional method of contraception is required for the pregnant partner.

Note: Abstinence is acceptable if this is the established and preferred contraception for the patient

Exclusion Criteria:

* Patients with a current diagnosis of diabetes mellitus are not eligible for this study.

Note: Patients with pre-diabetes or previous diabetes or glucose intolerance and who are currently not taking any diabetes medications are eligible

* Patients taking medications that cannot be safely stopped during the fasting periods or which may not be safely taken without food are not eligible for this study
* Received prior systemic cytotoxic chemotherapy, biological therapy, radiotherapy, or major surgery within 3 weeks prior to first dose of study drug. A 1-week washout is permitted for palliative radiation to non-central nervous system (CNS) disease, with approval from the principal investigator
* History of syncope with caloric restriction or another medical comorbidity which would make fasting potentially dangerous
* Current use of oral vitamin C supplements
* Currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigation device within 3 weeks of first dose of current study drug
* Expected to require any other form of systemic or localized antineoplastic therapy while on trial (including maintenance therapy with another agent, radiation therapy, and/or surgical resection)
* History of anti-PD1 or anti-CTLA4 therapy
* Unresolved toxicity ≥ CTCAE grade 2 except for neuropathy, alopecia
* Untreated brain or leptomeningeal metastases or previously treated CNS metastases with any of the following: residual neurologic deficit; history of seizures; ongoing requirement of steroids, exceeding prednisone 10 mg daily dose
* Patients who have uncontrolled or severe hyponatremia, hypernatremia, syndrome of inappropriate antidiuretic hormone secretion (SIADH), hypokalemia, hyperkalemia, hypomagnesemia, or hypermagnesemia
* Patients who have glucose-6-phosphate dehydrogenase (G6PD) deficiency, hereditary spherocytosis, or other conditions predisposing patient to hemolysis
* Patients who have a history of oxalate renal calculi
* Major surgery within 4 weeks of first dose of immunotherapy
* Known severe (grade ≥ 3) hypersensitivity reactions to fully human monoclonal antibodies, antibody, or severe reaction to immuno-oncology agents, such as colitis or pneumonitis requiring treatment with steroids; or has a history of interstitial lung disease, any history of anaphylaxis, or uncontrolled asthma
* Evidence of bleeding diathesis or clinically significant coagulopathy
* Receiving systemic corticosteroid therapy 1 week prior to the first dose of study drug or receiving any other form of systemic immunosuppressive medication.

Note: Corticosteroid use as a premedication for IV contrast allergies/reactions is allowed. Patients who are receiving daily corticosteroid replacement therapy are also an exception to this rule. Daily prednisone at doses of ≤ 10 mg or equivalent hydrocortisone dose are examples of permitted replacement therapy. Use of inhaled or topical corticosteroid is permitted

* Active or history of autoimmune disease that requires systemic treatment within 2 years of the start of study drug (i.e., use of disease-modifying agents, corticosteroids, or immunosuppressive drugs).

Note: Patients with autoimmune conditions requiring hormone replacement therapy or topical treatments are eligible

* Has had an allogeneic tissue/solid organ transplant, except for corneal transplants
* Legally incapacitated or has limited legal capacity
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, active coronary artery disease, myocardial infarction or cerebrovascular accident within 6 months prior to study entry, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2027-01-15 (Estimated); Study Completion 2028-01-15 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who adhere to the fast mimicking diet | Up to 30 months
  Adherence will be defined as the percentage of patients who adhere to the fasting-mimicking diet ≥ 75% of the designated days and receive all doses of study drugs for at least any 2 cycles of therapy during the course of the study. Adherence will be reported overall and by cycle started.
Incidence of adverse events (AEs) | Up to 30 months
  The frequency and severity of treatment-related events will be assessed using Common Terminology Criteria for Adverse Events version 5.0. Descriptive statistics will be used to summarize AEs including counts for categorical measures and means for continuous measures. Incidence of AEs will be reported overall and by cycle started.

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to 30 months
  ORR will be evaluated using Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1. Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm; Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters; Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions); Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Progression-free survival (PFS) | Up to 30 months
  Measured from start of treatment to the date of event defined as the first documented progression or death due to any cause. PFS Progression will be evaluated using RECIST v1.1. Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions).
Overall survival (OS) | Up to 30 months
  Measured from start of treatment until death from any cause. Patients who are still alive at the time of the analysis, or who have become lost to follow-up or withdrawn consent will be censored at their last date known to be alive.

CONTACTS AND LOCATIONS:
Overall Officials: Diana Hanna, MD, Principal Investigator — University of Southern California
Locations (2):
- United States (2):
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California